CLINICAL TRIAL: NCT04889079
Title: Assessing Adolescent Use of Nexplanon Over Time: a Prospective, Longitudinal Study
Brief Title: Assessing Adolescent Use of Nexplanon Over Time
Status: Active, not recruiting | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Rebecca Simmons, Principal Investigator, University of Utah
Other Study IDs: IRB_00142231
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Contraception
Keywords: adolescents; contraception; contraceptive implant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adolescent females, aged 15-18: Adolescents females aged 15-18, who selected a contraceptive implant to prevent pregnancy.
  Interventions: Behavioral: Contraceptive use (continuation/switching/discontinuation)
- Adolescent females, aged 19-24: Adolescents females aged 19-24, who selected a contraceptive implant to prevent pregnancy.
  Interventions: Behavioral: Contraceptive use (continuation/switching/discontinuation)

INTERVENTIONS:
Behavioral: Contraceptive use (continuation/switching/discontinuation) — Assessing contraceptive continuation/switching/discontinuation over 12-months

SUMMARY:
The purpose of this study is to compare Nexplanon decision-making, uptake, satisfaction and contraceptive outcomes (continuation, switching, discontinuation) over a 12-month period among adolescents ages 15-18 to adolescents ages 19-24, living in Utah. Data from this study will provide valuable information for clinical and public health offerings, counseling and support for Nexplanon use across stages of adolescence.

DETAILED DESCRIPTION:
Despite increasing availability of Nexplanon in the United States, only limited resesarch exists on Nexplanon use among adolescents, particularly nulliparous adolescents. A Cochrane systematic review of long-acting contraception use among adolescents in 2017 identified only four studies that had specifically assessed implant use and continuation among adolescents [1]. Of these, the majority of studies assessed use postpartum [1]. The majority of research on adolescent attitudes around and barriers to long-acting reversible contraception has been conducted on intrauterine devices, rather than implants, and further research is needed to understand decision-making and behaviors around implant use [2]. Additionally, no studies have assessed differences in adolescent decision-making by age. While adolescence is considered ages 10-24 [3], this period is one of substantial change, physically, mentally, and in stages of life. Contraceptive use can be influenced by all of these [4] and understanding differences in stages of adolescence could result in meaningful differences in counseling and support approaches.

The purpose of this study is to compare Nexplanon decision-making, uptake, satisfaction and contraceptive outcomes (continuation, switching, discontinuation) over a 12-month period among adolescents ages 15-18 to adolescents ages 19-24, living in Utah. Data from this study will provide valuable information for clinical and public health offerings, counseling and support for Nexplanon use across stages of adolescence.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 15-24;
* Not currently pregnant;
* Planning to avoid pregnancy for the next 12 months;
* Selecting the contraceptive implant as their contraceptive method of choice;
* Willing to be contacted via email survey 4 times over 12-months

Exclusion Criteria:

-

Ages: 15 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Adolescents living in Utah seeking a contraceptive implant at a participating clinic.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Estimated)
Dates: Start 2021-06-06 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
12-month contraceptive outcomes | 12-months
  This outcome measures contraceptive use. The question asks "are you still using the Nexplanon implant that you received", and then the outcomes are either: continuation, switching or discontinuation.

SECONDARY OUTCOMES:
Contraceptive satisfaction | 12-months
  The 5-point Likert satisfaction scale asks "how satisfied are you with your Nexplanon implant?" and the scale ranges from 1-Very unsatisfied to 5-Very satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Berlan ED, Richards MJ, Vieira CS, Creinin MD, Kaunitz AM, Fraser IS, Edelman A, Mansour D. Best Practices for Counseling Adolescents about the Etonogestrel Implant. J Pediatr Adolesc Gynecol. 2020 Oct;33(5):448-454. doi: 10.1016/j.jpag.2020.06.022. Epub 2020 Jul 2. PMID 32621879
- [Background] Sawyer SM, Azzopardi PS, Wickremarathne D, Patton GC. The age of adolescence. Lancet Child Adolesc Health. 2018 Mar;2(3):223-228. doi: 10.1016/S2352-4642(18)30022-1. Epub 2018 Jan 30. PMID 30169257
- [Background] Downey MM, Arteaga S, Villasenor E, Gomez AM. More Than a Destination: Contraceptive Decision Making as a Journey. Womens Health Issues. 2017 Sep-Oct;27(5):539-545. doi: 10.1016/j.whi.2017.03.004. Epub 2017 Apr 12. PMID 28412049
- [Result] Diedrich JT, Klein DA, Peipert JF. Long-acting reversible contraception in adolescents: a systematic review and meta-analysis. Am J Obstet Gynecol. 2017 Apr;216(4):364.e1-364.e12. doi: 10.1016/j.ajog.2016.12.024. Epub 2016 Dec 28. PMID 28038902